CLINICAL TRIAL: NCT01631838
Title: Effects of Tocotrienols Supplementation on Platelet Aggregation in Subjects With Metabolic Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malaysia Palm Oil Board (Other Government)
Collaborators: Universiti Putra Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: PD157/11
Record Dates: First submitted 2012-06-26; First posted 2012-06-29 (Estimated); Last update posted 2013-12-20 (Estimated); Status verified 2013-12

CONDITIONS: Metabolic Syndrome; Platelet Aggregation, Spontaneous
Keywords: Tocotrienols; Platelet aggregation; Metabolic syndrome; Platelet activation; Thrombosis
MeSH Terms: conditions — Metabolic Syndrome; Platelet Aggregation, Spontaneous; Thrombosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tocotrienol-rich fraction 400mg (Experimental)
  Interventions: Dietary Supplement: Tocotrienol-rich fraction 400mg
- Placebo (Experimental)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Tocotrienol-rich fraction 400mg — Tocovid Suprabio 200mg is taken twice daily (after breakfast and dinner) for 2 weeks. During postprandial day (Day 14), subjects are requested to consume breakfast meal containing 50g of fat and 100mL of milkshake, follow by capsule consumption
  Other Names: TOCOVID SupraBio 200mg
  Arms: Tocotrienol-rich fraction 400mg
Dietary Supplement: Placebo — Placebo is taken twice daily (after breakfast and dinner) for 2 weeks. During postprandial day (Day 14), subjects are requested to consume breakfast meal containing 50g of fat and 100mL of milkshake, follow by capsule consumption
  Other Names: Palm Olein
  Arms: Placebo

SUMMARY:
The objective of this study is to address the anti-thrombotic effects of tocotrienols supplementation via modulation of platelet activation, thrombotic markers, inflammatory markers and endothelial function.

It is hypothesized that 2 weeks supplementation of tocotrienols will be able to suppress platelet aggregation in subjects with metabolic syndrome.

DETAILED DESCRIPTION:
A double-blind, randomized, crossover study comparing the effects of tocotrienols vs. placebo will be conducted in subjects with metabolic syndrome. Subjects will be supplemented with Tocovid Suprabio 200 mg twice daily (or placebo) for 2 weeks followed by a postprandial challenge on Day 14. During the postprandial challenge, venous blood samples will be collected during fasting. Subjects are then required to consume a high fat breakfast meal containing 50g fat and 100mL milkshake, followed by the assigned capsules. Venous blood samples will be drawn at 2, 4 and 6 hours after consumption of capsules. A washout period of at least 14 days will be in place before the commencement of the second treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 25-60 year
* Haemoglobin level >11.5 g/dL in women and >12.5 g/dL in men
* Serum ferritin > 15µg/L
* According to Clinical Practice Guidelines, Management of Type 2 Diabetes Mellitus in Malaysia (2009), metabolic syndrome subjects are identified with:
* Waist circumference ≥ 90 cm in men and ≥ 80 cm in women

and with any two of the following criteria:

* Elevated triacylglycerols > 1.7 mmol/L
* Low HDL cholesterol < 1.0 mmol/L in men and < 1.3 mmol/L in women
* Elevated blood pressure ≥ 130/≥85 mm Hg
* Fasting glucose ≥ 5.6 mmol/L to 7 mmol/L

Exclusion Criteria:

* Medical history of myocardial infarction, angina, ischemic attack, hemorrhagic stroke, deep vein thrombosis, coronary artery disease, bleeding disorder, cancer, allergy to vitamin E
* Smoker
* Lactose intolerance
* Pregnancy or lactation
* Current use of vitamin E, medications modulating blood coagulation, hypertension, lipid-lowering and glucose-lowering agents, corticosteroids
* Significant hepatic and renal impairment
* Fever, cold or infection during bleeding day
* Alcoholic

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2012-05; Primary Completion 2012-08 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Platelet Aggregation | Day 0 - fasting, Day 14 - fasting, Day 14 - 4hr
  Comparison will be made between Day 14-fasting and changes will be measured between Day 14-fasting and 4hr.

SECONDARY OUTCOMES:
Platelet activation | Day 0 - fasting, Day 14 - fasting, Day 14 - 4hr
  Comparison will be made between Day 14-fasting and changes will be measured between Day 14-fasting and 4hr.
Haemostatic markers (Plasminogen activator inhibitor type 1 and sP-selectin) | Day 0 - fasting, Day 14 - fasting, Day 14 - 2hr, Day 14 - 4hr, Day 14 - 6 hr
  Comparison will be made between Day 14-fasting and postprandial response will be compared between two interventions
Inflammatory markers (sE-selectin, sICAM-1, and sVCAM-1) | Day 0 - fasting, Day 14 - fasting, Day 14 - 4hr
  Comparison will be made between Day 14-fasting and postprandial response will be compared between two interventions
Lipid Profile | Day 0 - fasting, Day 14 - fasting
  Comparison will be made between Day 14-fasting
D-dimer | Day 0 - fasting, Day 14 - fasting, Day 14 - 4hr
  Comparison will be made between Day 14-fasting and postprandial response will be compared between two interventions
Full blood count and liver function test | Day 0-fasting and Day 14-fasting
  Comparison will be made between Day 14-fasting

CONTACTS AND LOCATIONS:
Overall Officials: Ju Yen Fu, PhD, Principal Investigator — Malaysia Palm Oil Board
Locations (1):
- Malaysia Palm Oil Board, Kajang, Selangor, Malaysia